CLINICAL TRIAL: NCT06129058
Title: Home-based Transcranial Direct Current Stimulation (tDCS) to Promote Social Communication and Behaviour in Children With Autism Spectrum Disorder (ASD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASDR02
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
Keywords: tDCS; MRI; brain stimulation
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomized sham-controlled
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and outcomes assessor will be blind to tDCS or sham condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (Experimental): active tDCS
  Interventions: Device: At-home transcranial direct current stimulation (tDCS)
- Sham (Sham Comparator): sham tDCS
  Interventions: Device: Sham at-home tDCS

INTERVENTIONS:
Device: At-home transcranial direct current stimulation (tDCS) — 30 minutes session 5 days/week for 3 weeks.
  Arms: tDCS
Device: Sham at-home tDCS — 30 minutes session 5 days/week for 3 weeks.
  Arms: Sham

SUMMARY:
Transcranial direct current stimulation (tDCS) is a form of non-invasive brain stimulation that can be delivered in a home setting. It is a safe and tolerable intervention that has shown promise for improving positive social communication and self-regulation in youth with Autism Spectrum Disorder (ASD). Children and youth with ASD will be randomized to At-home tDCS or sham control stimulation for 3 weeks. We will measure the effect of At-home tDCS on the brain mechanisms and clinical measures of social communication and self-regulation..

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a form of non-invasive brain stimulation that can be delivered in a home setting. It is a safe and tolerable intervention that has shown promise for improving positive social communication and self-regulation in youth with Autism Spectrum Disorder (ASD). Previous studies have been limited by small and poorly represented samples, lack of experimental control, insufficient follow-up periods, inadequate blinding and the absence of neural outcome measures. Our project will collect pilot data on the effects of home-based tDCS on reducing disruptive behaviours in youth with ASD, in order to inform the design of a follow-up full-scale clinical trial. We will recruit youth with ASD who experience clinically significant difficulties with social communication and self-regulation. Participants will be randomized to tDCS or sham control stimulation for 3 weeks. We will measure the effect of tDCS on the brain mechanisms and clinical measures of social communication and self-regulation..

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of autism spectrum disorder and self-regulation impairment or social communication challenges
* Able to participate in tDCS

Exclusion Criteria:

* Children with contraindications to tDCS (history of seizures, family history of seizures, metal implants)
* Co-existing neurological conditions (epilepsy, stroke, etc.)

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment | weeks 1-18
  Recruitment rates of 4 participants/month are achieved with a ≥ 20% response rate
Attrition | weeks 1-18
  Attrition rates of less than 10% (i.e., ≥90% of participants successfully complete assessments).
Adherence | weeks 1-18
  90% of participants who complete assessment achieve the target intensity and dose (15 tDCS sessions)
Blinding | weeks 1-18
  Blinding of participants and their parents/caregivers and required study team using a Blinding Questionnaire indicating the perceived group membershipmembers will be assessed using a Blinding Questionnaire indicating the perceived group membership (tDCS/Sham)

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | 0 weeks, 6 weeks, 18 weeks
  Diffusion imaging - change in fractional anisotropy, Resting State functional MRI change in Blood Oxygen Level Dependent (BOLD) signal
Inhibitory control | 0 weeks, 6 weeks, 18 weeks
  change in Go/No Task Response Time
Overall Clinical Change | 0 weeks, 6 weeks, 18 weeks
  Clinical Global Impression scale - 1 item on a scale from 0-7 (a change of 0.5 indicates a clinical impact of significance)

CONTACTS AND LOCATIONS:
Locations (1):
- Holland Bloorview Kids Rehabilitation Hosptail, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbo N, Mitchell T, Tonekaboni SH, Anagnostou E, Andrade BF, Thorpe K, Beal DS. Feasibility and usability of remote transcranial direct current stimulation (tDCS) for self-regulation in children with autism: protocol for a randomized controlled pilot study. Pilot Feasibility Stud. 2025 Apr 29;11(1):57. doi: 10.1186/s40814-025-01650-4. PMID 40301914